CLINICAL TRIAL: NCT07048379
Title: Comparison of Orthotics, Physical Therapy, and Physical Therapy+Orthotics in Patients With Carpal Tunnel Syndrome
Brief Title: Different Treatment Approaches for Carpal Tunnel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Emel Tasvuran, PhD; Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 254
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Orthotic Devices; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Orthosis (Experimental): Participants will be given a rest orthosis for 3 weeks.
  Interventions: Device: Orthosis
- Physical Therapy (Experimental): Participants will receive physical therapy treatment for 3 weeks (15 sessions). Each physical therapy session will consist of hot packs and TENS applications, tendon-nerve sliding exercises, stretching and strengthening exercises.
  Interventions: Other: Physical Therapy
- Orthosis+Physical Therapy (Experimental): Both orthotic and physical therapy interventions will be applied for 3 weeks.
  Interventions: Device: Orthosis; Other: Physical Therapy

INTERVENTIONS:
Device: Orthosis — A resting orthosis will be preferred because it keeps the wrist in a neutral position.
  Other Names: 3 weeks
  Arms: Orthosis; Orthosis+Physical Therapy
Other: Physical Therapy — Participants will undergo physical therapy for three weeks, including hot packs, TENS, tendon-nerve sliding exercises, stretching and strengthening exercises.
  Arms: Orthosis+Physical Therapy; Physical Therapy

SUMMARY:
Carpal tunnel syndrome is a common syndrome in the upper extremities resulting from compression of the median nerve, which branches out to the first three fingers of the wrist. The project will be studied in three separate groups. The first group consists of patients who only use orthoses, the second group consists of patients who only receive physical therapy, and the third group consists of patients who receive both orthoses and physical therapy. The aim of all three groups is to examine the effects of the interventions on the daily living activities, pain, grip strength, and quality of life of patients with carpal tunnel syndrome and to evaluate the patients' satisfaction levels after the interventions. As part of the study, the group using orthoses will be given a resting orthosis that keeps the wrist in a neutral position. The group receiving physical therapy will be administered Transcutaneous Electrical Nerve Stimulation (TENS) current, hot packs, and exercises. The third group will receive both the orthosis approach and the physical therapy approach. Ultimately, this project aims to help determine the most beneficial intervention for patients with carpal tunnel syndrome by comparing these three interventions.

DETAILED DESCRIPTION:
Carpal tunnel syndrome is a peripheral neuropathy caused by compression of the median nerve in the wrist. It is a syndrome that is commonly seen in approximately 1-5% of the population throughout their lifetime. It is more common in middle-aged women. Conservative treatment is generally preferred for mild to moderate carpal tunnel syndrome. Conservative treatment allows for the reduction or even elimination of symptoms associated with this syndrome without the need for surgery. Individuals can continue their daily lives as usual. The use of orthoses, one of these methods, plays an important role in the treatment of carpal tunnel syndrome. Orthotics minimise movement of the wrist, preventing compression in this area, contributing to functional improvement and benefiting the individual's daily activities. Using orthotics throughout the day can have a positive effect on the individual's condition by reducing and preventing inflammation of the median nerve. Another conservative treatment approach is physical therapy. In physical therapy, exercises to strengthen the wrist muscles, stretching exercises to increase joint range of motion, and hot-cold applications in people with carpal tunnel syndrome are also effective in reducing pain. Additionally, there are patients who use orthoses and undergo physical therapy. When comparing the treatment periods of this group of patients to the other two groups, it is believed that their recovery periods will be shorter and they will recover more quickly than with the other two approaches. This study's aim is investigating the effects of the three intervention approaches on patients' quality of life, daily living activities, reduction in pain intensity, and grip strength, taking patient satisfaction into account. The project will be examined across three separate groups. The first group consists of patients who use only orthoses, the second group consists of patients who receive only physical therapy, and the third group consists of patients who receive both orthoses and physical therapy. The aim of all three groups is to examine the effects of the interventions on the daily living activities, pain, grip strength, and quality of life of patients with carpal tunnel syndrome and to evaluate the patients' satisfaction levels after the interventions. As part of the study, the group using orthoses will be given a resting orthosis that keeps the wrist in a neutral position. The group receiving physical therapy will be administered Transcutaneous Electrical Nerve Stimulation (TENS) current, hot packs, and exercises. The third group will receive both the orthosis approach and the physical therapy approach. Ultimately, this project aims to help determine the most beneficial intervention for patients with carpal tunnel syndrome by comparing these three interventions.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 65
* Have been diagnosed with mild or moderate carpal tunnel syndrome

Exclusion Criteria:

* Symptom duration of more than 12 months,
* Those who have undergone surgery for carpal tunnel syndrome
* Those who have received physical therapy within the last 6 months,
* Those who have received steroid injections into the carpal tunnel,
* Those with a history of trauma to the wrist and surrounding area,
* Those using non-steroidal anti-inflammatory drugs,
* Individuals with additional systemic, musculoskeletal, or neurological conditions that may affect symptoms will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Pain (visual analogue scale) | Pain will be assessed before and immediately after the interventions (3 weeks later).
  Pain will be assessed using a visual analogue scale. "Zero point" means that there is no pain and "Ten point" is unbearable pain according to scale.

CONTACTS AND LOCATIONS:
Overall Officials: Emel TAŞVURAN HORATA, Principal Investigator — Sakarya University of Applied Sciences; Gizem Nur ÇALIŞIR, Study Chair — Sakarya University of Applied Sciences; Nimet UÇAROĞLU CAN, Study Chair — Sakarya University; Sinem AKTAŞ, Study Chair — Sakarya University of Applied Sciences; Tülay KARSLI, Study Chair — Sakarya University of Applied Sciences; Ayşenur Yaren BÜRTEK, Study Chair — Sakarya University of Applied Sciences; Emre Uzun, Study Chair — Sakarya University

IPD SHARING:
Plan to Share IPD: No